CLINICAL TRIAL: NCT03546725
Title: The Effect of Compression Stockings on Edema and Discomfort During Short Haul Flights: A Randomized Controlled Trial
Brief Title: The Effect of Compression Stockings on Edema and Discomfort During Short Haul Flights
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Joachim Hjalde Halmsted Olsen, Bachelor of Medical Science, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 8392100
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Edema Leg
MeSH Terms: interventions — Stockings, Compression

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to wear a compression stocking on either the left or the right leg during a 3 - 3.5 hour flight. All participants will act as their own control, and as a result all data will be paired.
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be self-reported, and the author that assesses the outcomes and performs data analyses will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leg with compression stocking (Experimental): Leg wearing compression stocking during the flight
  Interventions: Device: Compression stocking
- Leg without compression stocking (No Intervention): Leg not wearing compression stocking during the flight

INTERVENTIONS:
Device: Compression stocking — Compression stocking with length below the knee and a class two compression level (corresponding to 23-32 mmHg compression).
  Arms: Leg with compression stocking

SUMMARY:
Compression stockings have beneficial effects on the development of venous thromboembolic complications and oedema during long- haul flights. A randomized controlled trial investigating the effect of compression stockings during short-haul flights with a duration less than fur ours is lacking. Deep vein thrombosis is very rare on flights shorter than four hours, but compression stocking could have beneficial effects on other outcomes. The aim of this study is to assess if compression stockings used during a 3-3.5-hour flight will decrease leg edema and discomfort.

DETAILED DESCRIPTION:
All participants will be adults who will undergo a 3-3.5 hours flight. Participants have received oral and written information about the trial. All compression stockings have a class two compression level (corresponding to 23-32 mmHg compression). Participants will be randomized to wear a compression stocking on one leg, while the other side acts as control. Within an hour preflight, the patient will measure ankle and calf circumference at marked circumferential areas on the leg and answer questionnaires regarding leg pain and subjective discomfort, whereafter the stocking will be put on, on the randomized side. Within one hour after the flight the stocking will be removed and patients will once again measure the ankle and calf circumference at the marked circumference and fill out the questionnaire.

Sample size: Mean difference in ankle circumference set to -0.19 cm. Standard deviation of the mean difference set to 0.3, 5% alfa and 80% power. Sample size with a paired design = at least 18 participants. However, for practical reasons we will include up to approximately 50 adults in the trial.

Withdrawal and dropout criteria: All participants can withdraw their consent at any point during the trial, without the need for explaining any reasons for withdrawal. Since compression stockings do not cause side effects, except for patients with severe arterial insufficiency in the legs, we do not expect the trial to be stopped due to complications. All withdrawals will be accounted for in the scientific publication.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥ 18 years of both sexes. Otherwise no restriction, since each participant acts as their own control.

Exclusion Criteria:

* Any condition requiring compression stockings during short-haul flights. Severe arterial insufficiency in the lower extremities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-05-26 (Actual); Study Completion 2018-05-26 (Actual)

PRIMARY OUTCOMES:
Ankle edema | Ankle circumference on the leg wearing a compression stocking and the leg not wearing compression stocking is measured up to one hour before, and one hour after flight.
  Difference in ankle circumference pre- and post flight on the leg with and the leg without compression stocking.

SECONDARY OUTCOMES:
Calf edema | Calf circumference on the leg wearing a compression stocking and the leg not wearing compression stocking is measured up to one hour before, and one hour after flight.
  Difference in calf circumference pre- and post flight on the leg with and the leg without compression stocking.
Leg pain | Leg pain is reported up to one hour before, and one hour after flight.
  Self-reported assessment of leg pain on a Visual Analogue Scale.
Leg discomfort | Leg discomfort is reported up to one hour before, and one hour after flight.
  Self-reported assessment of leg discomfort on a Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim HH Olsen, BScMed, Principal Investigator — Center for Perioperative Optimisation, Department of Surgery, Herlev og Gentofte Hospital, University of Copenhagen; Stina Öberg, MD, Study Director — Center for Perioperative Optimisation, Department of Surgery, Herlev og Gentofte Hospital, University of Copenhagen; Jacob Rosenberg, MD, DMSc, Study Director — Center for Perioperative Optimisation, Department of Surgery, Herlev og Gentofte Hospital, University of Copenhagen
Locations (1):
- Center for Perioperative Optimisation, Department of Surgery, Herlev og Gentofte Hospital, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olsen JHH, Oberg S, Rosenberg J. The effect of compression stocking on leg edema and discomfort during a 3-hour flight: A randomized controlled trial. Eur J Intern Med. 2019 Apr;62:54-57. doi: 10.1016/j.ejim.2019.01.013. Epub 2019 Feb 7. PMID 30738701